CLINICAL TRIAL: NCT05796960
Title: European Multicenter Study on Perioperative Management, Operative Strategy, Morbidity, and Outcomes of the Surgical Management of Advanced Thyroid Cancer: (EUROCRINE® Study Group).
Brief Title: European Multicenter Study on Surgical Management of Advanced Thyroid Cancer
Acronym: ATCEU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4999
Record Dates: First submitted 2023-03-16; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Thyroid Carcinoma; Thyroid Cancer; Thyroid Neoplasms; Thyroid Cancer, Papillary; Thyroid Cancer, Follicular; Thyroid Medullary Carcinoma; Anaplastic Thyroid Cancer
Keywords: Thyroid carcinoma; Eurocrine; Surgical management; Stage IV
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary; Thyroid cancer, follicular; Carcinoma, Medullary; Thyroid Carcinoma, Anaplastic | interventions — Thyroidectomy; Lymph Node Excision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical operations for advanced thyroid cancer: All adult (18 years old and older) patients registered in EUROCRINE® database with stage IV thyroid cancer, M1, N1b, or T3b and above will be included
  Interventions: Procedure: Thyroidectomy with or without lymphadenectomy or multivisceral resection

INTERVENTIONS:
Procedure: Thyroidectomy with or without lymphadenectomy or multivisceral resection — Lymph node dissection, as well as its surgical extension, was performed according to the surgeon's discretion. Multivisceral operations involved oesophagus, trachea and larynx.

SUMMARY:
The main aim of the study is to evaluate peri-operative surgical characteristics, operation extent, postoperative morbidity, and outcomes in patients undergoing surgery for advanced thyroid cancer in different European centers using the EUROCRINE® database.

DETAILED DESCRIPTION:
The incidence of thyroid cancer has risen exponentially over the last decades among developed countries. Even though this is mainly attributed to small well differentiated carcinomas (DTC) with excellent prognosis, the rates of advanced disease have also elevated. While the characteristics of advanced thyroid cancer are intuitively recognized by experienced surgeons of the field, a common definition among scientific societies is yet to be reached. The four main features of advanced cancer are locally and regionally advanced disease, distant metastasis, and recurrence. Guidelines for the optimal treatment of advanced disease are mainly included in the broader guidelines of each cancer subtype, such as the American Thyroid Association (ATA) guidelines for DTC, Medullary Thyroid Carcinoma (MTC) and most recently Anaplastic Thyroid Carcinoma (ATC). In the European setting, the European Society for Medical Oncology (ESMO) 2019 guidelines on thyroid cancer include a subsection for the management of advanced disease of each thyroid cancer type. A common limitation among published guidelines is the moderate to low level of evidence upon which the advanced disease recommendations are based; however, broad consensus has been reached regarding the paramount importance of surgery if an R0/R1 resection is achievable. Recently, new advances in targeted therapy guided by genetic alterations found in the tumor have provided new treatment options for patients; therefore, latest guidelines encourage the inclusion of patients with advanced disease in these clinical trials. Finally, neoadjuvant therapy modalities are constantly gaining ground with promising results allowing a greater portion of patients to benefit from surgery.

ELIGIBILITY:
Inclusion Criteria:

* All adult (18 years old and older) patients
* underwent surgery
* final histology of advanced thyroid carcinoma
* among European centers that participate in the Eurocrine® database between 2015 and 2021

Exclusion Criteria:

* Patients <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with final histology of advanced thyroid carcinoma operated among European centers that participate in the Eurocrine® database between 2015 and 2021
Sampling Method: Non-Probability Sample
Enrollment: 3917 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Perioperative characteristics | January 2015-January 2021
  Descriptive analysis of surgical perioperative characteristics of patients undergoing surgery for advanced thyroid cancer in European centers.

SECONDARY OUTCOMES:
Short-term clinical outcomes | January 2015-January 2021
  Descriptive analysis of short-term clinical outcomes of patients undergoing surgery for advanced thyroid cancer in European centers in terms of RLN palsy, critical neurovascular injury and voice changes through otorhinolaryngologist and clinical post-operative evaluation
Short-term clinical outcomes | January 2015-January 2021
  Descriptive analysis of short-term clinical outcomes of patients undergoing surgery for advanced thyroid cancer in European centers in terms of surgical complications, such as bleeding, lymphorrea tracheal or oesophageal injury (detected through clinical and/or imaging evaluation).
Short-term clinical outcomes | January 2015-January 2021
  Descriptive analysis of short-term clinical outcomes of patients undergoing surgery for advanced thyroid cancer in European centers in terms of hypocalcemia, hypoparathormonemia (detected through clinical and/or laburatoristic evaluation).

OTHER OUTCOMES:
Overall survival, recurrence and mortality | January 2015-January 2021
  Descriptive analysis of overall survival, recurrence and mortality in patients undergoing surgery for advanced thyroid cancer in European centers.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Raffaelli, Prof, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Reasonable requests will be evaluated by the Eurocrine Council